CLINICAL TRIAL: NCT02509650
Title: Identification of Mutations Responsible for Rare Familial Skin Diseases by Next Generation Sequencing
Acronym: DERMA-SEQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6024
Record Dates: First submitted 2015-07-15; First posted 2015-07-28 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Familial Lipomatosis; Very Rare Dermatologic Diseases
Keywords: Exome sequencing; Skin disease; Familial lipomatosis
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of the protocol is to use next generation sequencing to identify pathogenic variants in genes involved in very rare skin diseases.

The secondary purpose will be to study the genotype-phenotype correlation in order to re-evaluate the classification of these disorders. This work could help in the understanding of the physiopathology of very rare skin disorders.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by familial lipomatosis
* patients with rare dermatologic disease without molecular diagnosis
* written informed consent is obtained from the patient and his/her family

Exclusion Criteria:

* the patient does not want to participate to the protocol
* the patient is already included in another study using next generation sequencing technologies

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Familial lipomatosis
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a deleterious mutation | 6 months
  Validation of the exome sequencing results will be done by sanger sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Salima EL CHEHADEH, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Fédération de Génétique, Service de Génétique Médicale, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de Dermatologie, Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg